CLINICAL TRIAL: NCT02609308
Title: Platelet Rich Plasma and Lateral Ankle Sprain. A Comparative Study
Brief Title: Lateral Ankle Sprain and Platelet Rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Nuevo Leon (Other)
Responsible Party: Principal Investigator, Carlos A Acosta-Olivo, MD, PhD, Universidad Autonoma de Nuevo Leon
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OR15-008
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2019-10-23 (Actual); Status verified 2019-09

CONDITIONS: Ankle Injuries
Keywords: ankle sprain; platelet-rich plasma; ankle injuries
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Use of platelet rich plasma in patients with ankle sprain
Who Masked: Investigator, Outcomes Assessor
Masking Description: Application of autologous platelet-rich plasma
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Short leg cast (Active Comparator): The patients in this group will be immobilize with a short leg cast for 14 days, and later they will be able to do physical rehabilitation and will be evaluated with American Orthopedic Foot and Ankle Society´s Ankle Hindfoot scale and Foot and Ankle Disability Index.
  Interventions: Other: Short leg cast
- Platelet-rich plasma (Experimental): In this group, the patients will be receive a single dose of autologous platelet-rich plasma, and will be immobilized with a short leg cast. Posteriorly, they will be evaluated with American Orthopedic Foot and Ankle Society´s Ankle Hindfoot scale and Foot and Ankle Disability Index.
  Interventions: Procedure: Platelet-rich plasma

INTERVENTIONS:
Other: Short leg cast — Immobilization with short leg cast with a dorsiflexed foot for two weeks
  Arms: Short leg cast
Procedure: Platelet-rich plasma — Will be applied 5 mL of autologous platelet-rich plasma under the lateral malleolus, over the anterior talofibular ligament
  Arms: Platelet-rich plasma

SUMMARY:
Lateral ankle sprains are one of the most common in sports medicine. Considering the sprains in general, they represent an 85% of the ankle lesions. The incidence in high performance athletes range from 16 to 21%. It is estimated that 10,000 to 25,000 peoples suffers a lateral ankle sprain per hour in the United States. The objective of the treatment is to normalize the articular function and allow the patient to return to his or her normal physical activities. Platelet rich plasma is a simple of autologous blood with concentrations of platelets above baseline values. This is rich in platelet derived growth factor which stimulates cell replication, angiogenesis, transforming growth factor B1, fibroblast growth factor, epidermal growth factor, and insulin like growth factor. The risks of its applications are minimal and are usually involved with allergic reactions to other medications that are applied in combination with the platelet-rich plasma.

To establish that the use of platelet rich plasma and immobilization with a short leg cast in acute lateral ankle sprains will enhance an early recovery in comparison with just immobilization with the cast.

DETAILED DESCRIPTION:
Lateral ankle sprains are one of the most common in sports medicine. Considering the sprains in general, they represent an 85% of the ankle lesions. The incidence in high performance athletes range form 16 to 21%. It is estimated that 10,000 to 25,000 suffers a lateral ankle sprain per hour in the United States. The objective of the treatment is to normalize the articular function and allow the patient to return to his or her normal physical activities.

The lateral ligamentous complex of the ankle consists of three ligaments: the anterior talofibular, the calcaneofibular, and the posterior talofibular. The anterior talofibular ligament is the most affected. The patient describes a tear sensation in the ankle after an acute inversion of it. The injuries occur during physical activities as running. The patients presents with pain, swelling and tenderness over the affected ligaments. The proper diagnosis of the sprain includes anteroposterior, lateral and mortise view X rays of the affected ankle; if there is any suspicion of instability of the ankle, the physician shall order a Magnetic Resonance Image (MRI) to evaluate the ligaments.

Lateral ankle sprains have been classified by numerous methods. By anatomic site, lateral ankle sprains can be classified as grade I: anterior talofibular sprain, grade II: anterior talofibular and calcaneofibular sprains, and grade III: anterior talofibular, calcaneofibular and posterior talofibular sprains. By clinical system the sprains can be classified as mild with minimal function loss, no limp, minimal swelling, tenderness, pain with reproduction of mechanism of injury; moderate with moderate functional loss, unable to rise on toes, limp when walking, localized swelling; and severe with diffuse tenderness, patient use crouches for ambulation.

Conventional treatment for lateral ankle sprains is conservative, but a 32% of the patients have chronic complications as edema, pain, and ankle instability. The treatment for acute sprains have good to excellent results. Ankle dorsiflexion allows the fibers of the affected ligament to approximate and gives stability of the ankle. The first phase of the treatment requires rest, immobilization, compression with orthesis, and the use of non steroidal anti-inflammatory drug.

Platelet rich plasma is a sample of autologous blood with concentrations of platelets above baseline values, is rich in platelet derived growth factor which stimulates cell replication, angiogenesis, transforming growth factor beta-1, fibroblast growth factor, epidermal growth factor, and insulin like growth factor. The risks of its applications are minimal and are usually involved with allergic reactions to other medications that are applied in combination with the platelet rich plasma.

Purpose To establish that the use of platelet rich plasma and immobilization with a short leg cast in acute lateral ankle sprains will enhance an early recovery in comparison with just immobilization with the cast.

ELIGIBILITY:
Inclusion Criteria:

* Acute lateral ankle sprain with no more of 48 hours of evolution
* First time lateral ankle sprain
* Grade 2 or 3

Exclusion Criteria:

* Associated pathologies like diabetes mellitus, osteoarthritis, rheumatoid arthritis, ankylosing spondylitis, neurologic or psychiatric issues
* Pregnant women
* Previous surgery of the foot and ankle
* Blood dyscrasias

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Acosta-Olivo, MD, PhD, Principal Investigator — Universidad Autonoma de Nuevo Leon
Locations (1):
- Universidad Autonoma de Nuevo Leon, Monterrey, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] van Dijk CN, Lim LS, Bossuyt PM, Marti RK. Physical examination is sufficient for the diagnosis of sprained ankles. J Bone Joint Surg Br. 1996 Nov;78(6):958-62. doi: 10.1302/0301-620x78b6.1283. PMID 8951015
- [Result] Anderson RB, Hunt KJ, McCormick JJ. Management of common sports-related injuries about the foot and ankle. J Am Acad Orthop Surg. 2010 Sep;18(9):546-56. doi: 10.5435/00124635-201009000-00006. PMID 20810936
- [Result] Bernuzzi G, Petraglia F, Pedrini MF, De Filippo M, Pogliacomi F, Verdano MA, Costantino C. Use of platelet-rich plasma in the care of sports injuries: our experience with ultrasound-guided injection. Blood Transfus. 2014 Jan;12 Suppl 1(Suppl 1):s229-34. doi: 10.2450/2013.0293-12. Epub 2013 Jul 3. PMID 23867186
- [Result] Frei R, Biosca FE, Handl M, Trc T. [Conservative treatment using plasma rich in growth factors (PRGF) for injury to the ligamentous complex of the ankle]. Acta Chir Orthop Traumatol Cech. 2008 Feb;75(1):28-33. Czech. PMID 18315959
- [Result] Hall MP, Band PA, Meislin RJ, Jazrawi LM, Cardone DA. Platelet-rich plasma: current concepts and application in sports medicine. J Am Acad Orthop Surg. 2009 Oct;17(10):602-8. doi: 10.5435/00124635-200910000-00002. PMID 19794217
- [Result] Halpern BC, Chaudhury S, Rodeo SA. The role of platelet-rich plasma in inducing musculoskeletal tissue healing. HSS J. 2012 Jul;8(2):137-45. doi: 10.1007/s11420-011-9239-7. Epub 2012 Jan 18. PMID 23874254
- [Result] Hammond JW, Hinton RY, Curl LA, Muriel JM, Lovering RM. Use of autologous platelet-rich plasma to treat muscle strain injuries. Am J Sports Med. 2009 Jun;37(6):1135-42. doi: 10.1177/0363546508330974. Epub 2009 Mar 12. PMID 19282509
- [Result] Petersen W, Rembitzki IV, Koppenburg AG, Ellermann A, Liebau C, Bruggemann GP, Best R. Treatment of acute ankle ligament injuries: a systematic review. Arch Orthop Trauma Surg. 2013 Aug;133(8):1129-41. doi: 10.1007/s00402-013-1742-5. Epub 2013 May 28. PMID 23712708
- [Derived] Blanco-Rivera J, Elizondo-Rodriguez J, Simental-Mendia M, Vilchez-Cavazos F, Pena-Martinez VM, Acosta-Olivo C. Treatment of lateral ankle sprain with platelet-rich plasma: A randomized clinical study. Foot Ankle Surg. 2020 Oct;26(7):750-754. doi: 10.1016/j.fas.2019.09.004. Epub 2019 Sep 28. PMID 31640921

RESULTS

PARTICIPANT FLOW:
Groups:
- Short Leg Cast: The patients in this group will be immobilize with a short leg cast for 14 days, and later they will be able to do physical rehabilitation and will be evaluated with American Orthopedic Foot and Ankle Society's Ankle Hindfoot scale and Foot and Ankle Disability Index.
  Short leg cast: Immobilization with short leg cast with a dorsiflexed foot for two weeks.
- Platelet-rich Plasma: In this group, the patients will be receive a single dose of autologous platelet-rich plasma, and will be immobilized with a short leg cast. Posteriorly, they will be evaluated with American Orthopedic Foot and Ankle Society's Ankle Hindfoot scale and Foot and Ankle Disability Index.
  Platelet-rich plasma: Will be applied 5 mL of autologous platelet-rich plasma under the lateral malleolus, over the anterior talofibular ligament.
Period: Overall Study
Arm/Group | Short Leg Cast | Platelet-rich Plasma
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Short Leg Cast | Platelet-rich Plasma | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.5 (15.4) | 27.9 (12.1) | 26.7 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 4 | 7 | 11
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 25.4 (3.8) | 26.8 (3.5) | 26.3 (3.6)
Visual Analog Scale (VAS) [Mean (Standard Deviation); unit: units on a scale] — The VAS assesses the pain level by assigning a score from 0 to 10, with 0 representing no pain and 10 representing the worst pain level.
  units on a scale | 8.0 (1.3) | 7.5 (1.9) | 7.8 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: American Orthopedic Foot and Ankle Society Ankle-Hindfoot Scale (AOFAS)
Description: Scale that evaluates pain, function and alignment of foot. The best score is 100 points, and the worst score are 0 points.
Time Frame: Sixth month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Short Leg Cast | Platelet-rich Plasma
Number analyzed (Participants) | 10 | 11
units on a scale | 97.8 (2.6) | 98.5 (3.4)

2. Secondary Outcome: Visual Analogue Scale
Description: Evaluate the pain in a scale of 0 to 10, when 0 is no pain, and 10 is the worst pain
Time Frame: Sixth month
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Short Leg Cast | Platelet-rich Plasma
Number analyzed (Participants) | 10 | 11
cm | 0.2 (0.40) | 0.1 (0.3)

3. Secondary Outcome: Foot and Ankle Disability Index (FADI)
Description: The Foot and Ankle Disability Index (FADI) assesses activities such as standing, walking on flat or uneven surfaces, walking on inclines, and the length of time of walking without difficulty. It also includes a section for sports activities and ankle or foot pain (or both). The highest score is 136 points, indicating the best clinical situation, free of pain and limitations, while the lowest score is 0.
Time Frame: Sixth month
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Short Leg Cast | Platelet-rich Plasma
Number analyzed (Participants) | 10 | 11
units on a scale | 135.3 (1.0) | 135.4 (1.0)

ADVERSE EVENTS:
Time Frame: All included patients were evaluated at 24 weeks after the protocol interventions were initiated.
Arm/Group | Short Leg Cast | Platelet-rich Plasma
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 0/11

LIMITATIONS AND CAVEATS:
The diagnosis of Lateral Ankle Sprain was based on a clinical classification. We didn't use an Ultrasound scan, to perform the application of the Platelet Rich Plasma, or to assess morphologically the affected area before and after the treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No